CLINICAL TRIAL: NCT04897906
Title: The Effect of Education Given to Primiparous Pregnant Women on Parental Self-Efficacy and Mother-Infant Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cisem Bastarcan, Research Assistant, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CBastarcan
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Pregnant Women
Keywords: Pregnancy; Mother-Infant Attachment; Parental Self-Efficacy; Education Pregnant

STUDY DESIGN:
Intervention Model Description: Pregnant women included in the research sample will be divided into two groups as experimental and control groups. Experimental group; is the group to be trained. Control group; It is the group in which no intervention will be made other than data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group; It is the group that will be given mother and neonatal care education.
  Interventions: Behavioral: Education Group
- Control Group (No Intervention): Control group; It is the group in which no intervention will be made other than data collection.

INTERVENTIONS:
Behavioral: Education Group — Mother care, newborn care and breastfeeding education will be provided to pregnant women in the third trimester of pregnancy.
  Arms: Experimental group

SUMMARY:
This research will be carried out in a quasi-experimental design to determine the effect of maternity care and neonatal care training given to primiparous pregnant women on parental self-efficacy and mother-infant attachment in the postpartum period.

Research Hypotheses:

H0: There is no difference in parental self-efficacy and mother-infant attachment in the postpartum period between pregnant women who received training during pregnancy and did not.

H1: There is a difference in parental self-efficacy and mother-infant attachment in the postpartum period between pregnant women who received and did not receive education during pregnancy.

DETAILED DESCRIPTION:
The number of people to be included in the study was made with the power analysis made considering the previous studies. With the G * Power (3.1.9.7.) Program, the number of samples for each group was determined as n = 34 at 80% power, 5% error and 95% confidence interval. Considering the losses in data collection, 20% was added to each group and it was decided to recruit a total of 80 people, 40 people for the experimental group and 40 people for the control group.

Pregnant women included in the research sample will be divided into two groups as experimental and control groups. Data will be collected by sending via an online questionnaire created by the researchers. Before the online questionnaire is sent to the experimental and control groups, the experimental-control days will be determined randomly by a lottery drawn by a third person (blinding). Pregnant women who agree to participate in the study will be assigned to the experimental and control groups according to the determined days.

The data obtained in the study will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Significance value will be considered as p <0.05.

Number, percentage, mean and standard deviation will be used as descriptive statistical methods in the evaluation of data. Pearson correlation and regression analysis will be applied among the continuous variables of the study. The t-test will be used to compare the quantitative continuous data between two independent groups, and the One-way Anova test will be used to compare the quantitative continuous data between more than two independent groups. After the Anova test, the Scheffe test will be used as a complementary post-hoc analysis to determine the differences.

ELIGIBILITY:
Inclusion Criteria:

* Being at 36-40 weeks of gestation
* Being her first pregnancy
* Being literate
* Being over the age of 18

Exclusion Criteria:

* Not in the 36-40 gestational week
* Not a first pregnancy
* Illiterate
* Under 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Parental self-efficacy in postpartum period of pregnant women who received education during pregnancy | Mothers will be evaluated within 30-40 days after birth.
  Parental Self-Efficacy Scale will be used in the evaluation. It is a scale developed to determine the personal beliefs of new parents about their competencies in their roles.
Mother-Infant attachment in postpartum period of pregnant women who received education during pregnancy | Mothers will be evaluated within 30-40 days after birth.
  Maternal Attachment Scale will be used in evaluation. It was developed to measure the mother's love and attachment to her baby. Higher scores on the scale indicate higher maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Cisem Bastarcan, MsC, Principal Investigator — Research Assistant
Locations (1):
- Beykent University, Büyükçekmece, Istanbul, Turkey (Türkiye)